CLINICAL TRIAL: NCT06407973
Title: A Randomized Clinical Trial of ab Interno Canaloplasty and Trabeculotomy With the OMNI Surgical System Compared to Standard Medical Treatment as a Standalone Procedure in Patients With Primary Open Angle Glaucoma
Brief Title: A Clinical Trial Comparing the OMNI Surgical System to Standard Medical Treatment in Patients With Primary Open Angle Glaucoma
Acronym: EVOLVE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision by the Sponsor
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09074
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost

STUDY DESIGN:
Intervention Model Description: Randomized controlled open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgical (OMNI Surgical System (OSS)) (Active Comparator): Canaloplasty followed by Trabeculotomy using the OMNI Surgical System.
  Interventions: Device: OMNI Surgical System
- Standard Medical Care (SMC) (Active Comparator): Standard Medical Care with Latanoprost and one or two adjunctive glaucoma medications at the discretion of the Principal Investigator
  Interventions: Drug: Latanoprost plus adjunctive glaucoma medication

INTERVENTIONS:
Device: OMNI Surgical System — The OMNI Surgical System is 510(k) cleared and indicated for canaloplasty (microcatheterization and transluminal viscodilation of Schlemm's canal) followed by trabeculotomy (cutting of trabecular meshwork) to reduce intraocular pressure in adult patients with primary open-angle glaucoma
  Other Names: OMNI
  Arms: Surgical (OMNI Surgical System (OSS))
Drug: Latanoprost plus adjunctive glaucoma medication — * Latanoprost ophthalmic solution (0.005%) is a topical prostaglandin F2 analog used in the treatment of Glaucoma.
  * Adjunctive topical glaucoma medication(s) as selected by the Investigator
  Arms: Standard Medical Care (SMC)

SUMMARY:
A Randomized Clinical Trial of Ab Interno Canaloplasty and Trabeculotomy with the OMNI® Surgical System Compared to Standard Medical Treatment as a Standalone Procedure in Patients with Primary Open Angle Glaucoma (EVOLVE)

DETAILED DESCRIPTION:
This prospective, multicenter, post-market clinical trial will evaluate the safety and effectiveness of canaloplasty and trabeculotomy using the OSS as a standalone procedure in patients with POAG.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 45 years or older.
2. History of uncomplicated cataract surgery and posterior chamber intraocular lens (IOL) implantation without compromise to the lens capsule, zonular dehiscence/rupture or vitreous prolapse, 6 months or more prior to Baseline Visit (pseudophakic subjects), OR, phakic and no anticipated need for cataract surgery over the study duration.
3. Under treatment with a topical prostaglandin F2 analog (e.g. latanoprost, travoprost, bimatoprost, tafluprost) either as monotherapy or in combination with one (1) adjunctive medication for a minimum of 6 weeks prior to the Screening visit.
4. Intraocular pressure (IOP) at the Screening visit of >18 and not exceeding 36 mmHg.
5. Diagnosed with primary open angle glaucoma (POAG).

Exclusion Criteria:

1. Any of the following prior ocular procedures:

   * Laser trabeculoplasty ≤180 days prior to baseline
   * Durysta ≤12 months prior to baseline unless failure is documented and topical medication including a prostaglandin analog is in use as per Inclusion criterion # 3.
   * Implanted with iStent (All types), Cypass, Xen, Express, glaucoma draining device/valve, or Hydrus Device; or
   * Prior canaloplasty, goniotomy, trabeculotomy, trabeculectomy, endoscopic cyclophotocoagulation (ECP), Cyclophotocoagulation or CPC (G probe)
   * Retinal laser procedure ≤3 months prior to baseline
2. Concurrent IOP-lowering procedure other than the study procedure (OSS) (e.g. ECP, CPC,etc.)
3. Forms of glaucoma other than POAG including but not limited to: Pigmentary, pseudoexfoliative, acute angle closure, normal tension, pre-perimetric, traumatic, congenital, malignant, uveitic, neovascular or severe glaucoma as documented in subject's medical record.
4. Women of childbearing potential if they are currently pregnant or intend to become pregnant during the study period; are breast-feeding; or are not in agreement to use adequate birth control methods to prevent pregnancy throughout the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Subjects with a ≥ 20% reduction | 12 months
  Proportion of subjects with a ≥ 20% reduction from medicated baseline in mean diurnal IOP (DIOP) at 12 months post-operatively

SECONDARY OUTCOMES:
Diurnal IOP (DIOP) between 6 and 18 mmHg (inclusive) | 12 months
  Proportion of eyes at 12 months post-randomization, with mean medicated diurnal IOP (DIOP) between 6 and 18 mmHg (inclusive).
Number of Ocular Hypotensive Medications | 12 months
  Mean number of ocular hypotensive medications used at 12 months
Tear break-up time (TBUT) | 12 months
  Proportion of eyes with a minimal clinically important difference (MCID) defined as a 1 category improvement, in tear beak-up time (TBUT)
Corneal or conjunctival staining | 12 months
  Proportion of eyes with improvement in corneal staining or conjunctival staining by at least one category with no worsening in either at 12 months compared to baseline.
OSDI score | 12 months
  Proportion of subjects with a MCID in ocular surface disease index (OSDI) score at 12 months compared to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - North Bay Eye Associates, Petaluma, California
  - University Eye Specialists, Maryville, Tennessee

IPD SHARING:
Plan to Share IPD: No